CLINICAL TRIAL: NCT05331066
Title: EXACT - Understanding immunE-related toXicities by multifACeT Profiling
Brief Title: Understanding immunE-related toXicities by multifACeT Profiling
Acronym: EXACT
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 5064
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A prospective observational cohort study of patients undergoing CPI therapy in which translational research is the fundamental aspect of the study.

DETAILED DESCRIPTION:
The study aims to enroll and obtain samples of investigational interest from 200 patients over a 36-month recruitment period. Blood and/ or stool samples will be taken at baseline, in context of irAE development / during CPI treatment and during follow-up. Skin samples may also be taken upon development of organspeciifc irAEs.

Further assessments at baseline or during the course of or following treatment will be conducted in accordance with standard institutional practice and will be clinically driven. Clinical data, samples and results from archival, current or prospective diagnostic or therapeutic procedures will be used for research purposes within EXACT.

IrAE clinical monitoring will be conducted in accordance with standard institutional practice and will be clinically driven.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18 years or older
* Confirmed diagnosis of any form of solid malignancy with a clinical indication and appropriate treatment plan to commence immune checkpoint inhibitor therapy

Exclusion Criteria:

* Medical or psychological condition that would preclude informed consent
* Planned participation in a drug trial receiving investigational agents
* Subjects who have previously commenced immune checkpoint inhibitor therapy prior to study entry.
* Subjects unable to comply with the study or sample schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to enroll and obtain samples of investigational interest from 200 patients with a confirmed diagnosis of any form of solid malignancy with a clinical indication and appropriate treatment plan to commence immune checkpoint inhibitor therapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2028-04-06 (Estimated); Study Completion 2028-04-06 (Estimated)

PRIMARY OUTCOMES:
Patients who experience irAEs | 36 months
  To determine the proportion of patients who experience irAEs during treatment with CPI.

SECONDARY OUTCOMES:
Biological and clinical characteristics | 60 months
  To profile biological and clinical characteristics at baseline and during treatment with CPI to detect indicators predictive of the development of immunotherapy-related adverse events (irAEs).
Time to development of irAEs | 36 months
  To determine time to clinical development of irAEs during treatment with CPI.
Proportion of patients experiencing irAEs | 60 months
  • To determine the proportion of patients experiencing any irAE during long-term follow up, post treatment.

OTHER OUTCOMES:
Impact on patients quality of life using patient questionnaires | 60 months
  • Explore the quality-of-life impact on patients enrolled in longitudinal multi-facet disease profiling and in patients who develop irAEs.

CONTACTS AND LOCATIONS:
Overall Officials: Samra Turajlic, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, Chelsea, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided